CLINICAL TRIAL: NCT06596447
Title: Neurophysiological Investigation of the Approach-avoidance Axis in OCD: Applications to Neuromodulation
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Nicole Provenza, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-56119
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Obsessive Compulsive Disorder (OCD); Neuromodulation
Keywords: Obsessive Compulsive Disorder; OCD; Deep Brain Stimulation; DBS
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with Treatment Resistance OCD
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — While most patients with obsessive compulsive disorder (OCD) eventually respond to treatment with medication and/or behavioral therapy, a small minority do not improve following all conventional treatments. Obsessive-compulsive disorder (OCD) can sometimes be difficult to treat with medication and psychotherapy. For these patients, in this study, we employ deep brain stimulation (DBS), an advanced surgical treatment that uses electrical impulses.

SUMMARY:
We will recruit 10 patients with OCD meeting established criteria for surgical evaluation. Following informed consent and baseline evaluations, each will be implanted with permanent DBS SenSight leads and the Medtronic Percept RC IPG, which has on-device neural recording capability and rechargeability.

We will collect a broad array of neurobehavioral data across two environments with complementary advantages: the clinic and the home. The first 2 Aims test our mechanistic hypothesis by studying the pattern of VS neural activity in the controlled environment of the lab/clinic during two complementary paradigms: one based on a psychophysical behavioral task, the other based on ERP, a therapeutic behavioral intervention. The third aim tests this hypothesis in an ambulatory, naturalistic setting with chronic neural on-device recordings paired with time resolved behavioral measures. We will investigate a possible common neural basis underlying approach and avoidance across these 3 paradigms.

Subjects will participate in research at 7 critical timepoints during routine clinic visits (Fig. 4): before implant, 1 day before DBS activation, immediately after DBS activation, 2 weeks, 3 months, 6 months, and 12 months after DBS initiation. At these timepoints, patients will complete clinical assessments, perform the Probabilistic Approach Avoidance Task (PAAT), and conduct exposure trials under the guidance of a psychologist. The clinic offers the most controlled environment and provides opportunities for collecting high temporal resolution behavior synchronized to local field potential (LFP) recordings. These data will allow us to identify the degree of overlap in the time-resolved neural activity driving individual decisions to approach potential rewards or avoid potential aversive stimuli (Aim 1), and resist performing compulsions in order to achieve relief after OCD symptoms are triggered (Aim 2).

At home, our goal is to investigate patient trajectories along the approach-avoidance axis as OCD symptoms improve (Aim 3). We will leverage passive, on device recordings that occur in the background of everyday life activities and synchronize these neural recordings with data collected via wearables, ecological assessments, and video diaries. Capturing neural and behavioral data in the home environment is essential for understanding the neural and behavioral changes that occur over longer timescales than individual clinical visits. The neurobehavioral biomarkers generated by this dataset will provide trackable readouts of clinical status that could inform therapeutic decision-making and enable data driven intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Principal diagnosis of OCD per DSM-5;
2. Adult between ages 18 and 64;
3. At least a five-year history of treatment-refractory OCD that causes substantial subjective distress and impairment in functioning;
4. Minimum score of 28 on the Y-BOCS;
5. Failed an adequate trial of at least three SSRIs;
6. Failed an adequate trial of clomipramine;
7. Failed augmentation of one or more of the aforementioned drugs with at least one anti-psychotic medication;
8. Failed an adequate trial of CBT for OCD, defined as 25 hours of documented exposure and response prevention (ERP) by an expert therapist;
9. Stable psychotropic medical regimen for the month preceding surgery;
10. Principal diagnosis of OCD who are approved by our multi-disciplinary team to undergo DBS surgery within two months of enrollment;
11. Ability to provide fully informed, written consent;
12. Availability of a family member or significant other who is willing to accompany patients to study visits if necessary.

Exclusion Criteria:

1. Lifetime diagnosis of psychotic disorder such as schizophrenia;
2. Alcohol or substance abuse/dependence within 6 months, excluding nicotine;
3. Concern for high risk of suicidal behavior or impulsivity;
4. Patient is [regnant or plans to become pregnant in the next 24 months;
5. Need for diathermy;
6. Existence of any neurological or medical condition/disorder that makes the individual, in the opinion of the study team, a poor candidate to participate in the intended study procedures
7. Comorbid psychiatric disorder that, in the opinion of the study team, may interfere with the candidate's ability to participate in study activities;
8. Primary diagnosis of a Hoarding Disorder.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study accepts individuals that are receiving DBS to treat OCD with a primary diagnosis of OCD and a 5-year history of treatment-refractory OCD.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Changes in OCD symptoms | 14 months
  Response will be defined as 35% decrease in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) from baseline. The range is from 0 to 40 with a score of 0-7 indicating subclinical symptoms, 8-15 mild symptoms, 16-23 moderate symptoms, 24-31 severe symptoms, and 32-40 extreme symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No